CLINICAL TRIAL: NCT02272569
Title: A Prospective, Non-comparative, Multi-center Clinical Trial to Evaluate the Safety and Efficacy of the STARflo Glaucoma Implant in Patients With Open Angle Glaucoma
Brief Title: STARflo European Safety and Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISM01
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Open Angle Glaucoma
Keywords: glaucoma; glaucoma drainage device; glaucoma shunt
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STARflo Glaucoma Implant (Experimental): Implantation of the STARflo Glaucoma Implant by an ab-externa technique with connection from the anterior chamber to the suprachoroidal space
  Interventions: Device: STARflo Glaucoma Implant

INTERVENTIONS:
Device: STARflo Glaucoma Implant — Implantation of the STARflo Glaucoma Implant following surgical technique described in European labelling. Procedure does not require the use of anti-fibrotic medications.

SUMMARY:
Prospective, Non-comparative, Multi-center clinical trial to evaluate the safety and efficacy of the STARflo Glaucoma Implant in patients with refractory open angle glaucoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter clinical trial to assess the efficacy and the safety of the STARflo™ Glaucoma Implant.

Patients will enter the study after providing written informed consent. Patients will be screened to confirm that they are eligible for study participation.

When eligibility has been established using the in/exclusion criteria, surgery will be scheduled.

Pre and post-surgery, patients will be evaluated at scheduled intervals (1 day, 1 week, 1 month, 3 months, 6 months, 12 months, 24 months) for a total duration of 24 months following surgery.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of refractory open angle glaucoma
* Documented 21 mmHg < IOP ≤ 40 mmHg, under medication
* Patient must provide written informed consent

Main Exclusion Criteria:

* Patients with diagnosis of glaucoma other than open angle glaucoma (e.g. angle closure glaucoma) in the study eye
* Patients who failed one or more cilio ablative procedure in the study eye if these cilio ablative procedures were performed as a consequence of previous failed filtering surgery
* Clinically significant intra-ocular inflammation or infection, presence of ocular disease such as uveitis, ocular infection, severe dry eye, severe blepharitis, active proliferative/inflammatory retinopathy in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Reduction in mean diurnal intraocular pressure (IOP) at 12 months vs. baseline IOP | 12 months
  IOP of each patients at baseline will be compared to IOP of patient after 12 months

SECONDARY OUTCOMES:
Reduction in mean diurnal intraocular pressure (IOP) at 24 months vs. baseline IOP | 24 months
  IOP of each patients at baseline will be compared to IOP of patient after 24 months
Reduction in number of IOP lowering medications at 12 months vs. baseline | 12 months
  compare number of active ingredient of each patients at baseline vs number of active ingredient after 12 months
Reduction in number of IOP lowering medications at 24 months vs. baseline | 24 months
  compare number of active ingredient of each patients at baseline vs number of active ingredient after 24 months
Rate of adverse events | 24 months
  assessment and counting of adverse events (% by adverse event) including procedure related complications
Visual Acuity | 12 months
  comparison of visual acuity at 12 months vs. baseline
Absolute success rate (%) at 12 months | 12 months
  absolute success: IOP < 21mmHg and < 5mmHg with a minimum of 30% IOP reduction compared to baseline without the need for concomitant glaucoma medication
Qualified success rate (%) at 12 months | 12 months
  qualified success: IOP < 21mmHg and < 5mmHg with a minimum of 30% IOP reduction compared to baseline with and without the need for concomitant glaucoma medication
Qualified success rate (%) at 24 months | 24 months
  qualified success: IOP < 21mmHg and < 5mmHg with a minimum of 30% IOP reduction compared to baseline with and without the need for concomitant glaucoma medication
Absolute success rate (%) at 24 months | 24 months
  absolute success: IOP < 21mmHg and < 5mmHg with a minimum of 30% IOP reduction compared to baseline without the need for concomitant glaucoma medication

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Chair — Sponsor Representative; Sheng Lim, Dr., Study Director — Medical Advisor
Locations (8):
- Belgium (2):
  - UZA, Edegem
  - CHU Sart Tilman, Liège
- MHAT Central Onco Hospital, Plovdiv, Bulgaria
- France (2):
  - Hopital de la Croix-Rousse, Lyon
  - CHNO des Quinze Vingts, Paris
- Germany (2):
  - University Clinic Heidelberg, Heidelberg
  - Ludwig-Maximilians-University Munich, Munich
- Universitatsklinik fur Augenheilkunde Inselspital, Bern, Switzerland